CLINICAL TRIAL: NCT07001813
Title: Clinical and Radiographic Assessment of the Outcomes of Dental Implant Inserted After Xenograft Socket Preservation in Posterior Maxilla: A Randomized Controlled Study
Brief Title: Clinical and Radiographic Assessment of the Outcomes of Dental Implant Inserted After Xenograft Socket Preservation in Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 545/2022
Record Dates: First submitted 2025-05-16; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Implant Therapy
Keywords: Implant; clinical stability; radiographic assessment; soft tissue health

STUDY DESIGN:
Intervention Model Description: This study was conducted on adults above the age of 21 years old with badly decayed posterior maxillary teeth (16 cases) requiring extraction, then subjected to implant placement. These patients were divided equally and http://www.randomizer.org randomly into two groups using Group (A) (8 cases): was treated by immediate socket preservation with S1-XB xenograft augmentation after extraction. Group (B) (8 cases): was not exposed to any type of socket preservation after the extraction procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket preserved (Active Comparator): (8 cases): was treated by immediate socket preservation with S1-XB xenograft augmentation after extraction.
  Interventions: Device: socket preserved
- non preserved sockets (Placebo Comparator): (8 cases): was not exposed to any type of socket preservation after the extraction procedure.
  Interventions: Device: non preserved socket

INTERVENTIONS:
Device: socket preserved — (8 cases): was treated by immediate socket preservation with S1-XB xenograft augmentation after extraction.
  Arms: socket preserved
Device: non preserved socket — (8 cases): was not exposed to any type of socket preservation after the extraction procedure.
  Arms: non preserved sockets

SUMMARY:
Clinical and Radiographic Assessment of the Outcomes of Dental Implant Inserted after Xenograft Socket Preservation in Posterior Maxilla: A Randomized Controlled Study

DETAILED DESCRIPTION:
Dental implants have become a common choice among the treatment options for missing teeth rehabilitation and has remarkably high survival and success rates Since the introduction of implants into clinical practice more than several decades ago. The success rate of dental implants, over the last ten years, has been about 90- 95%.

Invasive and non-invasive clinical tests are available like histomorphometric analysis, radiographic analysis, push- and pull-out tests, percussion tests, Periotest and resonance frequency analysis (RFA) are employed to assess the steadiness of dental implants to assess objectively implant stability at different stages of its service life to verify successful implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 21 and 40 years.
* General good health.
* Absence of any relevant systemic disease.
* Presence of a hopeless maxillary posterior tooth that requires extraction.
* Extraction site suitable for replacement by a dental implant.
* Cases have adequate bone width and length.
* Volunteer subjects must sign an informed consent.

Exclusion Criteria:

* Poor oral hygiene with no possibility of improvement.
* Smokers (more than 10 cigarettes per day).
* Chronic treatment with any medication known to affect oral status and bone turnover.
* Drug or alcohol abuse.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — males with general good health.
Enrollment: 16 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
clinical assessment of primary stability of dental implant | immediately and after four months • A ratchet was used to place the implant immediately The implant stability using OSTELL device was taken immediately postoperative implant insertion and was assessed after 4 months before prothesis
  implant stability assessment by
  1. rachet insertion torque
     * The implant was installed into the osteotomy site using the motorized method with the engine set at 50 rpm and 35-50 N/cm torque.
     * A ratchet was used to place the implant to the desired depth when the insertion torque was more than 35N/cm torque.
  2. osstell device (ISQ) Make it possible to monitor osseointegration in a precise and objective manner.
     * Osstell helps to objectively and non-invasively determine implant stability. The prob attached to the instrument via a cable and measurements are displayed on the black lit display.
     * The device held in a right angle to the center toward the implant to be examined, the maximum deviation angle from the orthoradial direction of percussion is 45 degrees. In addition, the rod and the test surface must maintain 0.6-2.5 mm distance according to the operating instructions.
     * The implant stability using OSTELL device was taken immediately postoperative and was assessed after 4 months
radiographic assessment of implant stability | 1.Pre-operative radiographic evaluation: before implant placement 2.Intra oral paralleling periapical direct digital radiographic procedure: immediately after placement and after four months
  1. Pre-operative radiographic evaluation:
     After a healing period of four months, all the patients evaluated by Scanora 3D Cone Beam Computed Tomography scanner (CBCT) for evaluation bucco-lingual dimention, mesio-distal width, relation to neighbouring vital structures, bone density and assessment good position for implant placement.
     Post-operative Digital Radiography Assessment:
  2. Intra oral paralleling periapical direct digital radiographic procedure:
  Indirect Standardized digital radiographs were achieved using KaVo Scan eXam™M One and the Rinn extension cone paralleling (XCP) periapical film holder. The KaVo Scan eXam™M One is an Intraoral digital imaging plate system (psp) system using Imaging plate which is a film-like thin, flexible, and wireless phosphorescent plate, which works as a wireless receptor.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed kamel Attia, postgraduate student, Principal Investigator — Suez Canal University
Locations (1):
- faculty of dentistry Suez canal university, Ismailia, Egypt

REFERENCES:
- [Background] AAl MA, El Far M, Sheta NM, Fayyad A, El Desouky E, Nabi NA, Ibrahim M. Correlation of Implant Stability Between Two Noninvasive Methods Using Submerged and Nonsubmerged Healing Protocols: A Randomized Clinical Trial. J Oral Implantol. 2020 Dec 1;46(6):571-579. doi: 10.1563/aaid-joi-D-19-00130. PMID 33494103